CLINICAL TRIAL: NCT01048788
Title: A Multicenter, Uncontrolled, Open-label Phase 3 Trial of OPC-41061 in Patients With Hepatic Edema - Investigation of the Safety of Treatment at 7.5 mg Beyond 7 Days and of the Effect of Dose Escalation to 15 mg
Brief Title: A Trial of OPC-41061 in Patients With Hepatic Edema - Investigation of the Safety of Treatment at 7.5 mg Beyond 7 Days and of the Effect of Dose Escalation to 15 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-08-002; JapicCTI-100983 (Registry Identifier: JAPIC)
Record Dates: First submitted 2010-01-07; First posted 2010-01-14 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; ascites; Tolvaptan; OPC-41061
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC (Experimental)
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061 — OPC-41061 tablets will be orally administered once daily after breakfast at 7.5 mg on Day 1 to 7 and at either 7.5 or 15 mg on Day 8 to 14.

SUMMARY:
OPC-41061 will be orally administered at 7.5 mg/day for 7 days to cirrhosis patients with ascites despite having received conventional diuretic therapy. Based on the change in body weight, on Day 7 it will be decided whether to continue administration at the same dose or to increase the dose, and then OPC-41061 will be orally administered for an additional 7 days at either 7.5 mg/day or, if diuretic effect for the initial 7-day administration is insufficient, at an increased dose of 15 mg/day. Plasma drug level, efficacy, and safety of OPC-41061 by 14-day repeated administration will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients judged as having cirrhosis* based on previous imaging diagnosis

  * Definition of cirrhosis includes patients with collateral circulation due to chronic hepatic impairment
* Patients with ascites in whom the dose of existing diuretics cannot be increased due to risk of adverse drug reactions such as electrolyte abnormalities, or in whom sufficient therapeutic effect cannot be obtained with existing diuretics
* Patients who have been receiving oral combination therapy with a loop diuretic and an anti-aldosterone agent from at least 7 days prior to receipt of informed consent, with a dose combination of either loop diuretic equivalent to furosemide 40 mg/day or higher plus spironolactone 25 mg/day or higher, or loop diuretic equivalent to furosemide 20 mg/day or higher plus spironolactone 50 mg/day or higher
* Patients who are hospitalized or who can be hospitalized for the trial
* Patients capable of giving informed consent
* Patients who, together with their partner, agree to use an appropriate method of contraception until 4 weeks after the final trial drug administration

Exclusion Criteria:

* Patients with any of the following complications or symptoms:
* Hepatic encephalopathy (hepatic coma of grade 2 or higher)
* Hepatocellular carcinoma with imaging-diagnosed vascular infiltration into trunk or primary branch of portal vein, inferior vena cava, or trunk of hepatic vein
* Endoscopic findings from screening examination or from within 30 days prior to screening examination indicating the need for new therapy for esophageal or gastric varices during the trial period
* Repeated hemorrhoidal bleeding due to rectal varicose veins within 30 days prior to informed consent
* Heart failure (New York Heart Association Class III or IV)
* Anuria
* Impaired urination due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
* Patients with a history of any of the following disorders:
* Cerebrovascular disorder within 30 days prior to informed consent
* Hypersensitivity or idiosyncratic reaction to benzazepine derivatives (such as mozavaptan hydrochloride or benazepril hydrochloride)
* Morbidly obese patients with a body mass index (BMI: body weight (kg)/height (m)2) exceeding 35
* Patients with sitting systolic blood pressure lower than 90 mmHg
* Patients with any of following abnormal clinical laboratory values at time of the screening examination: Hemoglobin lower than 8.0 g/dL, total bilirubin higher than 4.0 mg/dL, serum creatinine higher than 2.0 mg/dL, serum sodium higher than 147 mEq/L, or serum potassium higher than 5.5 mEq/L
* Patients who are unable to take oral medication
* Female patients who are pregnant, possibly pregnant, or breast-feeding, or who are planning to become pregnant
* Patients who have used albumin preparations (therapeutic agents for hypoalbuminemia) or blood products containing albumin from within 7 days prior to informed consent
* Patients who received any investigational drug other than OPC-41061 within 30 days prior to informed consent
* Patients who have previously received OPC-41061
* Any patient who, in the opinion of the principle investigator or subinvestigator, is inappropriate for participation in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Chubu Region
  - Chugoku Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Discontinued/Terminated Before Day8: Subjects who disconrinued treatment before Day 7 or terminated by meeting the criteria on Day 7
- Continued Administration at 7.5 mg/Day: Subjects who did not meet the criteria for dose escalation
- Dose Escalation to 15 mg/Day: Subjects who met the criteria for dose escalation
Period: Overall Study
Arm/Group | Discontinued/Terminated Before Day8 | Continued Administration at 7.5 mg/Day | Dose Escalation to 15 mg/Day
Started | 8 | 30 | 13
Completed | 3 | 28 | 11
Not Completed | 5 | 2 | 2
Not completed — Adverse Event | 5 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Discontinued/Terminated Before Day8 | Continued Administration at 7.5 mg/Day | Dose Escalation to 15 mg/Day | Total
Number analyzed (Participants) | 8 | 30 | 13 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (6.8) | 63.9 (8.2) | 61.0 (11.4) | 63.5 (8.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 14 | 8 | 26
  >=65 years | 4 | 16 | 5 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 4 | 15
  Male | 6 | 21 | 9 | 36
Region of Enrollment [Number; unit: participants]
  Japan | 8 | 30 | 13 | 51

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Changes in body weight from baseline at the end of administration
Time Frame: Baseline, Day 14 or end of administration
Measure: Mean (Standard Deviation); unit: Kg
Groups:
- Discontitued/Terminated Before Day 8: Subjects who discontinued treatment before Day 7 or teiminated by meeting the criteria on Day 7
Arm/Group | Discontitued/Terminated Before Day 8 | Continued Administration at 7.5 mg/Day | Dose Escalation to 15 mg/Day
Number analyzed (Participants) | 8 | 30 | 13
Kg | -0.76 (0.93) | -2.97 (2.57) | -0.05 (2.30)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Discontinued/Terminated Before Day8 | Continued Administration at 7.5 mg/Day | Dose Escalation to 15 mg/Day
Serious Adverse Events (participants affected / at risk) | 3/8 | 3/30 | 2/13
Other Adverse Events (participants affected / at risk) | 7/8 | 22/30 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discontinued/Terminated Before Day8 (N=8) | Continued Administration at 7.5 mg/Day (N=30) | Dose Escalation to 15 mg/Day (N=13)
Positional Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia Obstructive (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septicaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Polyneuropathy Alcoholic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discontinued/Terminated Before Day8 (N=8) | Continued Administration at 7.5 mg/Day (N=30) | Dose Escalation to 15 mg/Day (N=13)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 2 (2)
Thirst (General disorders) | 1 (1) | 10 (10) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 4 (5) | 0 (0)
Blood Pressure Decreased (Investigations) | 1 (1) | 3 (4) | 1 (1)
Blood Urea Increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 2 (2)
Bladder Dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No